CLINICAL TRIAL: NCT04355741
Title: Gut Microbiota, "Spark and Flame" of COVID-19 Disease
Status: Completed | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Hospital de São Francisco Xavier, Centro Hospitalar de Lisboa Ocidental (Unknown); Centro Hospitalar Universitário São João (Unknown); CUF Academic and Research Medical Center (Unknown); Hospital CUF Infante Santo, S.A. (Unknown); Centro de Medicina Laboratorial Germano de Sousa, S.A. (Unknown); CINTESIS - Center for Health Technology and Services Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVID19_Microbiota
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: COVID-19; Gut microbiota
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ambulatory: Patients that are self-isolated at home
  Interventions: Other: Exposure
- Ward: Patients that are in an isolated room at the hospital
  Interventions: Other: Exposure
- ICU: Patients that are in the ICU of the hospital
  Interventions: Other: Exposure

INTERVENTIONS:
Other: Exposure — Individuals with SARS-CoV-2 exposure and COVID-19 symptoms.

SUMMARY:
Elderly, hypertension, diabetes and cardiovascular diseases are risk factors for COVID-19 morbility and mortality. However, the real reason for this is not yet understood. It is well documented that gut microbiota has a critical role in health, particularly in the immune system and therefore, we propose that gut microbiota composition could affect vulnerability and disease outcomes of COVID-19.

DETAILED DESCRIPTION:
In order to explore this hypothesis, we will analyse the gut microbiota of SARSCoV-2 infected patients categorized according to location: [1] ambulatory (self-isolation at home), [2] ward and [1] ICU; and severity.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years and above.
* COVID-19 patients.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients admitted to Portuguese hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Differences in gut microbiota composition between COVID-19 patients with different degrees of disease severity. | Stool samples of COVID-19 patients will be collected after subject enrollment (single point collection)

SECONDARY OUTCOMES:
Differences in gut microbiota composition between COVID-19 patients in relation to mortality. | Through study completion, an average of 3 months.
Differences in gut microbiota composition between COVID-19 patients in relation to length of stay in hospitals. | Through study completion, an average of 3 months.
Differences in gut microbiota composition between COVID-19 patients in relation to duration of mechanical ventilation. | Through study completion, an average of 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — Universidade Nova de Lisboa; Pedro Póvoa, PhD, Principal Investigator — Hospital São Francisco Xavier; Cristina Granja, PhD, Principal Investigator — Centro Hospitalar Universitário São João; Maria JR Sousa, PhD, Principal Investigator — Centro de Medicina Laboratorial Germano de Sousa, S.A.; José Leal, PhD, Study Chair — Centro de Medicina Laboratorial Germano de Sousa, S.A.
Locations (3):
- Portugal (3):
  - Hospital CUF Infante Santo, S.A., Lisbon
  - Hospital de São Francisco Xavier, Lisbon
  - Centro Hospitalar Universitário São João, Porto

IPD SHARING:
Plan to Share IPD: No